CLINICAL TRIAL: NCT06080178
Title: Goal-directed Fluid Therapy During Deep Inferior Epigastric Perforator (DIEP) Free Flap Breast Reconstruction - a Randomised Controlled Trial
Brief Title: Goal-directed Fluid Therapy During Deep Inferior Epigastric Perforator (DIEP) Free Flap Breast Reconstruction
Acronym: GDFT DIEP-flap
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Silvie Allaert, Principal Investigator, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMS.2023.036
Record Dates: First submitted 2023-09-22; First posted 2023-10-12 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hypotension During Surgery
Keywords: arterial hypotension; postoperative hypotension; Goal-directed Fluid Therapy; DIEP free flap breast reconstruction
MeSH Terms: conditions — Hypotension | interventions — Plasma-lyte 148; Norepinephrine

STUDY DESIGN:
Intervention Model Description: A monocentric, prospective, non-inferiority, randomised controlled trial. Interventional, phase IV trial. Patients will be randomly assigned to either a static intraoperative fluid management (reflecting the current standard of care), with a limitation of 5ml/kg/h crystalloids from induction of anaesthesia to completed skin closure, or a dynamic goal-directed fluid management, where crystalloid fluids are only administered during surgery if PPV is above 12%.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static group (Active Comparator): When during surgery systolic blood pressure (SBP) is below 100mmHg:
  * give a fluid bolus (Plasmalyte A) until 5ml/kg/h crystalloid (without maintenance infusion) is reached or until SBP is above 100mmHg
  * if the 5ml/kg/h crystalloid limit is already reached: start or increase norepinephrine infusion until SBP is above 100mmHg (with a maximum dose of 0.2mcg/kg/min).
  When SBP is above 120mmHg: decrease the norepinephrine infusion rate until SBP is below 120mmHg.
  When SBP remains below 100mmHg after reaching a vasopressor dose of 0.2mcg/kg/min: the anaesthetist can decide to give a bolus of 6mg ephedrine intravenous (IV) (with a maximum dose of 12mg ephedrine iv per hour).
  Interventions: Drug: Plasma-lyte (static group); Drug: Norepinephrine (static group)
- Dynamic group (Experimental): After insertion of an arterial line, a pulse contour analysis system will be installed (Acumen IQ sensor, Edwards) for measuring PPV and cardiac index (CI).
  When during surgery SBP is below 100mmHg and PPV is above 12%:
  • give a fluid bolus (Plasmalyte A) until PPV is below or equal to 12% or SBP is above 100mmHg
  When during surgery SBP is below 100mmHg and PPV is below or equal to 12%:
  • start or increase norepinephrine infusion until SBP is above 100mmHg (with a maximum dose of 0.2mcg/kg/min) When SBP is above 120mmHg: decrease the norepinephrine infusion rate until SBP is below 120mmHg.
  When SBP remains below 100mmHg after reaching a vasopressor dose of 0.2mcg/kg/min, and CI is < 2.2 L/min/m², a bolus of 6mg ephedrine iv will be given (with a maximum dose of 12mg ephedrine iv per hour).
  Interventions: Drug: Plasma-lyte (dynamic group); Drug: Norepinephrine (dynamic group)

INTERVENTIONS:
Drug: Plasma-lyte (static group) — Plasmalyte will be administered intravenously: (1) as a maintenance infusion 1ml/kg/h (from anaesthesia induction until ICU/PACU discharge); (2) as a fluid bolus until 5ml/kg/h crystalloid (without maintenance infusion) is reached or until SBP is above 100mmHg
  Arms: Static group
Drug: Norepinephrine (static group) — When during surgery SBP is below 100mmHg, if the 5ml/kg/h crystalloid limit is already reached, start or increase norepinephrine infusion until SBP is above 100mmHg (with a maximum dose of 0.2mcg/kg/min).
  Arms: Static group
Drug: Plasma-lyte (dynamic group) — Plasmalyte will be administered intravenously:
  (1) as a maintenance infusion 1 ml/kg/h (from anaesthesia induction until ICU/PACU discharge); (2) as a fluid bolus until PPV is below or equal to 12% or SBP is above 100mmHg.
  Arms: Dynamic group
Drug: Norepinephrine (dynamic group) — When during surgery SBP is below 100mmHg and PPV is below or equal to 12%: start or increase norepinephrine infusion until SBP is above 100mmHg (with a maximum dose of 0.2mcg/kg/min).
  When SBP is above 120mmHg: decrease the norepinephrine infusion rate until SBP is below 120mmHg.
  Arms: Dynamic group

SUMMARY:
Adequate free flap perfusion during Deep Inferior Epigastric Perforator (DIEP) flap breast reconstruction surgery requires maintaining blood pressure above 100 mmHg and avoiding excessive fluid administration. This study aims to determine whether the use of a measurement of preload dependency (Pulse Pressure Variation = PPV), can guide fluid therapy and if it decreases the risk of flap oedema. For this purpose, two fluid management strategies will be compared:

* Static intraoperative fluid management: Administration of crystalloid fluids is limited to 5ml/kg/h
* Dynamic intraoperative fluid management: Crystalloid fluids are only administered if PPV exceeds 12% The purpose of this study is to compare the static and dynamic (= targeted) fluid strategy and to evaluate the effect on flap oedema and flap perfusion.

DETAILED DESCRIPTION:
For adequate free flap perfusion during Deep Inferior Epigastric Perforator (DIEP) flap breast reconstruction surgery, blood pressure must remain sufficiently high. General anaesthesia often induces systemic hypotension. To counteract this hypotension, the anaesthetist administers intravenous fluids (crystalloid fluids). However, fluid overload can lead to an increased risk of flap oedema and decreased flap perfusion and in exceptional cases to flap failure. To maintain blood pressure above 100 mmHg and to avoid excessive fluid administration, a vasopressor (norepinephrine) can be administered. This reduces the amount of fluids administered, thereby reducing the risk of flap oedema.

This study aims to determine whether the use of a measurement of preload dependency (Pulse Pressure Variation = PPV), can guide fluid therapy and if it decreases the risk of flap oedema. To this end, two fluid management strategies will be compared:

* Static intraoperative fluid management: Administration of crystalloid fluids is limited to 5ml/kg/h
* Dynamic intraoperative fluid management: Crystalloid fluids are only administered if PPV exceeds 12% The purpose of this study is to compare the static and dynamic (= targeted) fluid strategy and to evaluate the effect on flap oedema and flap perfusion.

All included patients are randomized in a 1:1 ratio to the static (n = 41) or dynamic group (n = 41).

To treat hypotension in patients randomized to the 'static' group, fluid administration is limited to 5 ml/kg/h. When the maximum fluid volume is administered but blood pressure remains below 100 mmHg, norepinephrine is administered.

Treatment of hypotension in patients randomized to the 'dynamic' (= targeted fluid therapy) group, is guided by PPV. PPV is measured continuously during the surgery and if the blood pressure is below 100 mmHg, fluids are only administered if PPV is > 12%. If blood pressure is below 100 mmHg but PPV is < 12% (indicating no fluid is needed), norepinephrine is administered.

At the end of the procedure, 2 sensors are applied, these sensors provide information about the perfusion of the free flap during patient's stay in Intensive Care or the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Female adult patients, between 18 and 70 years of age
* Patients scheduled for DIEP free flap breast reconstruction
* Signed written informed consent form (ICF)

Exclusion Criteria:

* present atrial fibrillation (AF)
* heart failure New York Heart Association (NYHA) classification 2 or higher
* chronic kidney disease (CKD) stage 3B or higher
* American Society of Anesthesiologists (ASA) classification III or higher
* known allergy to study specific medication
* participation in another clinical trial
* Inability of the patient to understand Dutch sufficiently
* Patients who are pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Total intraoperative fluid volume | From anaesthesia induction until completed skin closure, assessed up to 12 hours
  Total intraoperative fluid volume (from anaesthesia induction until completed skin closure)

SECONDARY OUTCOMES:
Cumulative perioperative fluid volume | From anaesthesia induction until ICU/ PACU discharge, assessed up to 72 hours
  Cumulative perioperative fluid volume (intraoperative fluid volume + fluid administered in the intensive care unit (ICU) or post-anaesthesia care unit (PACU))
Cumulative perioperative norepinephrine dose | From anaesthesia induction until ICU/ PACU discharge, assessed up to 72 hours
  Cumulative perioperative norepinephrine dose (intraoperative and postoperative norepinephrine dose)
Peri- and postoperative blood lactate levels | From anaesthesia induction until ICU/ PACU discharge, assessed up to 72 hours
  Peri- and postoperative blood lactate levels (hourly measurement during surgery, every four hours in the ICU until discharge)
Percentage of time Systolic Blood Pressure (SBP) was above 100mmHg | During surgery, from anaesthesia induction until completed skin closure, assessed up to 12 hours
  Percentage of time SBP was above 100mmHg during surgery
Postoperative free flap tissue oxygenation and blood perfusion (tissue oximetry) | From ICU admission until ICU/ PACU discharge, assessed up to 60 hours
  Postoperative free flap perfusion monitored by near-infrared spectroscopy (NIRS) during ICU/PACU stay
Surgical complications | At ICU/ PACU discharge, assessed up to 60 hours and at hospital discharge, assessed up to 2 weeks
  Surgical complications (e.g. total or partial flap loss, venous flap congestion, hematoma) assessed at ICU/PACU discharge and at hospital discharge
Length of stay | From ICU admission until ICU/ PACU discharge, assessed up to 60 hours
  ICU/PACU length of stay (LOS) (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Silvie Allaert, MD, Principal Investigator — AZ Maria Middelares Gent
Locations (1):
- AZ Maria Middelares, Ghent, East Flanders, Belgium